CLINICAL TRIAL: NCT02839343
Title: Preoperative Extended Chemotherapy vs. Chemotherapy Plus Hypofractionated Radiation Therapy for Borderline Resectable Adenocarcinoma of the Head of the Pancreas
Brief Title: Combination Chemotherapy With or Without Hypofractionated Radiation Therapy Before Surgery in Treating Patients With Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Sky Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A021501; NCI-2016-00456 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2016-07-14; First posted 2016-07-20 (Estimated); Results first posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-04

CONDITIONS: Pancreatic Adenocarcinoma; Borderline Resectable Adenocarcinoma of the Head of the Pancrease
MeSH Terms: interventions — Radiotherapy; Surgical Procedures, Operative; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mFOLFIRINOX + surgery + FOLFOX (Experimental): Patients receive 8 cycles of mFOLFIRINOX. One cycle is 14 days. mFOLFIRINOX consists of oxaliplatin, irinotecan, leucovorin and 5-FU. Patients undergo surgery and receive 4 cycles of FOLFOX 4-12 weeks after surgery. FOLFOX consists of oxaliplatin, leucovorin and 5-FU.
  Interventions: Procedure: surgery; Drug: mFOLFIRINOX; Drug: FOLFOX
- mFOLFIRINOX + radiation + surgery + FOLFOX (Experimental): Patients receive 7 cycles of mFOLFIRINOX. One cycle is 14 days. mFOLFIRINOX consists of oxaliplatin, irinotecan, leucovorin and 5-FU. Patients receive radiation therapy then undergo surgery and receive 4 cycles of FOLFOX 4-12 weeks after surgery. FOLFOX consists of oxaliplatin, leucovorin and 5-FU.
  Interventions: Radiation: radiation therapy; Procedure: surgery; Drug: mFOLFIRINOX; Drug: FOLFOX

INTERVENTIONS:
Radiation: radiation therapy
  Arms: mFOLFIRINOX + radiation + surgery + FOLFOX
Procedure: surgery
Drug: mFOLFIRINOX — oxaliplatin IV, irinotecan IV, leucovorin IV and 5-FU IV
Drug: FOLFOX — oxaliplatin IV, leucovorin IV and 5-FU IV

SUMMARY:
This randomized phase II trial studies how well combination chemotherapy (mFOLFIRINOX) with or without hypofractionated radiation therapy before surgery works in patients with pancreatic cancer that can be removed by surgery. Drugs used in combination chemotherapy, such as oxaliplatin, leucovorin calcium, fluorouracil, and irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. It is not yet known if combination chemotherapy is more effective with or without hypofractionated radiation therapy before surgery in treating patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate and estimate 18 months overall survival (OS) rate of patients with borderline resectable pancreatic ductal adenocarcinoma (PDAC) receiving neoadjuvant therapy.

SECONDARY OBJECTIVES:

I. To evaluate and estimate the R0 resection rates in patients receiving each of the two multimodality treatment regimens.

II. To evaluate and estimate the event-free survival in patients receiving each of the two multimodality treatment regimens.

III. To evaluate and estimate the pathologic compete response (pCR) rates in patients receiving each of the two multimodality treatment regimens.

IV. To assess the adverse events (AE) profile and safety of each treatment arm.

TERTIARY OBJECTIVES:

I. To test the effect of the rs2853564 vitamin D receptor (VDR) variant on OS rate and discover novel candidate genes associated with OS and severe toxicity of chemotherapy by using genome-wide genotyping approaches.

II. To evaluate risk classification previously developed by Koay et al using normalized area under the enhancement curve (NAUC).

III. To access prognostic value of NAUC ratio defined as post-neoadjuvant NAUC divided by pre-neoadjuvant therapy NAUC.

IV. To evaluate risk classification previously developed by Koay et al using delta measure.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive oxaliplatin intravenously (IV) over 2 hours, irinotecan IV over 90 minutes, and leucovorin calcium IV over 2 hours on day 1. Patients also receive fluorouracil IV continuously over 46-48 hours on days 1-2. Treatment repeats every 14 days for 8 courses in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive oxaliplatin intravenously (IV) over 2 hours, irinotecan IV over 90 minutes, and leucovorin calcium IV over 2 hours on day 1. Patients also receive fluorouracil IV continuously over 46-48 hours on days 1-2. Treatment repeats every 14 days for 7 courses in the absence of disease progression or unacceptable toxicity. Patients receive either stereotactic body radiation therapy (SBRT) or hypofractionated image guided radiation therapy (HIGRT) on days 1-5 of course 8.

SURGERY Within 4 to 8 weeks after the last dose of chemotherapy (arm A) or of radiation (arm B), patients considered surgical candidates for resection (after central review) will undergo surgery at the registering institution.

ADJUVANT CHEMOTHERAPY Within 4-12 weeks from the date of surgery, patients will receive oxaliplatin IV over 2 hours and leucovorin IV over 2 hours on day 1. Patients also receive fluorouracil IV continuously over 46-48 hours on days 1-2. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 16 weeks for 2 years, then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of radiographic stage as borderline resectable disease by real-time Alliance central radiographic review
* No prior chemotherapy or radiation for pancreatic cancer
* No definitive resection of pancreatic cancer
* Chronic concomitant treatment with strong inhibitors of cytochrome p450, family 3, subfamily a, polypeptide 4 gene (CYP3A4) is not allowed on this study; patients on strong CYP3A4 inhibitors must discontinue the drug for 14 days prior to registration on the study
* Chronic concomitant treatment with strong CYP3A4 inducers is not allowed; patients must discontinue the drug 14 days prior to the start of study treatment
* No grade >= 2 neuropathy
* No known Gilbert's syndrome or known homozygosity for UGAT1A1*28 polymorphism
* No uncontrolled gastric ulcer disease (grade 3 gastric ulcer disease) within 28 days of registration
* Not pregnant and not nursing; for women of childbearing potential only, a negative pregnancy test done =< 7 days prior to registration is required
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine =< 1.5 x upper limit of normal (ULN) or
* Calculated (calc.) creatinine clearance > 45 mL/min
* Total bilirubin =< 2.0 mg/dL
* Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) =< 2.5 X upper limit of normal (ULN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Katz, MD, FACS, Study Chair — M.D. Anderson Cancer Center
Locations (155):
- United States (154):
  - Southern Cancer Center PC-Mobile, Mobile, Alabama
  - Southern Cancer Center PC-Springhill, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - University Oncology Associates, Clovis, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Saint Agnes Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Lincoln/LCI-Lincoln, Charlotte, North Carolina
  - Levine Cancer Institute-SouthPark, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Mallard Creek, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - NHRMC Radiation Oncology - Supply, Supply, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - NHRMC Radiation Oncology - 16th Street, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - IMG Hematology Oncology 8501, Fairfax, Virginia
  - IMG Hematology Oncology 8505, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Snyder RA, Zemla TJ, Shi Q, Segovia D, Ahmad SA, O'Reilly EM, Herman JM, Katz MHG. Postoperative Adverse Events Following Neoadjuvant Therapy and Surgery for Borderline Resectable Pancreatic Cancer in a Phase 2 Clinical Trial (Alliance A021501). Ann Surg Oncol. 2024 Oct;31(10):7033-7042. doi: 10.1245/s10434-024-15670-6. Epub 2024 Jul 15. PMID 39008208
- [Derived] Katz MHG, Shi Q, Meyers J, Herman JM, Chuong M, Wolpin BM, Ahmad S, Marsh R, Schwartz L, Behr S, Frankel WL, Collisson E, Leenstra J, Williams TM, Vaccaro G, Venook A, Meyerhardt JA, O'Reilly EM. Efficacy of Preoperative mFOLFIRINOX vs mFOLFIRINOX Plus Hypofractionated Radiotherapy for Borderline Resectable Adenocarcinoma of the Pancreas: The A021501 Phase 2 Randomized Clinical Trial. JAMA Oncol. 2022 Sep 1;8(9):1263-1270. doi: 10.1001/jamaoncol.2022.2319. PMID 35834226
- [Derived] Katz MHG, Ou FS, Herman JM, Ahmad SA, Wolpin B, Marsh R, Behr S, Shi Q, Chuong M, Schwartz LH, Frankel W, Collisson E, Koay EJ, Hubbard JM, Leenstra JL, Meyerhardt J, O'Reilly E; Alliance for Clinical Trials on Oncology. Alliance for clinical trials in oncology (ALLIANCE) trial A021501: preoperative extended chemotherapy vs. chemotherapy plus hypofractionated radiation therapy for borderline resectable adenocarcinoma of the head of the pancreas. BMC Cancer. 2017 Jul 27;17(1):505. doi: 10.1186/s12885-017-3441-z. PMID 28750659

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 (mFOLFIRINOX + Surgery + FOLFOX): Patients receive 8 cycles of mFOLFIRINOX. One cycle is 14 days. mFOLFIRINOX consists of oxaliplatin, irinotecan, leucovorin and 5-FU. Patients undergo surgery and receive 4 cycles of FOLFOX 4-12 weeks after surgery. FOLFOX consists of oxaliplatin, leucovorin and 5-FU.
- Arm 2 (mFOLFIRINOX + Radiation + Surgery + FOLFOXx): Patients receive 7 cycles of mFOLFIRINOX. One cycle is 14 days. mFOLFIRINOX consists of oxaliplatin, irinotecan, leucovorin and 5-FU. Patients receive radiation therapy then undergo surgery and receive 4 cycles of FOLFOX 4-12 weeks after surgery. FOLFOX consists of oxaliplatin, leucovorin and 5-FU.
Period: Overall Study
Arm/Group | Arm 1 (mFOLFIRINOX + Surgery + FOLFOX) | Arm 2 (mFOLFIRINOX + Radiation + Surgery + FOLFOXx)
Started | 70 | 56
Completed | 65 | 55
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Disease Progression Prior to Treatment | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (mFOLFIRINOX + Surgery + FOLFOX) | Arm 2 (mFOLFIRINOX + Radiation + Surgery + FOLFOXx) | Total
Number analyzed (Participants) | 70 | 56 | 126
Age, Continuous [Median (Full Range); unit: years] | 63 [37 to 83] | 66.5 [40 to 80] | 64 [37 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 28 | 62
  Male | 36 | 28 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 2 | 5
  White | 59 | 51 | 110
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Rate
Description: Defined as the percentage of patients who are alive at 18 months after randomization divided by the total number of evaluable patients in each arm. An evaluable patient is defined as any patient who signed informed consent, deemed eligible by central review and received any protocol-defined treatment. 95% confidence interval will be estimated based on standard method. Chi-squared test (or Fisher's exact test if the data in contingency table is sparse) will be used to compare 18 month OS rates among treatment arms. OS within each arm will be summarized by Kaplan-Meier method. Median, 1-year and 2-year rates will be estimated based on Kaplan-Meier curves.
Time Frame: 18 months
Population: Excluded from analysis were 6 patients that withdrew or progressed prior to treatment.
Measure: Number; unit: percentage of patients
Arm/Group | Arm 1 (mFOLFIRINOX + Surgery + FOLFOX) | Arm 2 (mFOLFIRINOX + Radiation + Surgery + FOLFOXx)
Number analyzed (Participants) | 65 | 55
percentage of patients | 64.6 | 47.3

2. Secondary Outcome: Residual Tumor (R)0 Resection Rate
Description: Defined as the percentage of patients in whom an achieved R0 resection was achieved during surgery.
Time Frame: 24 months
Population: Excluded from analysis were 6 patients that withdrew or progressed prior to treatment.
Measure: Number; unit: percentage of patients
Arm/Group | Arm 1 (mFOLFIRINOX + Surgery + FOLFOX) | Arm 2 (mFOLFIRINOX + Radiation + Surgery + FOLFOXx)
Number analyzed (Participants) | 65 | 55
percentage of patients | 49 | 35

3. Secondary Outcome: Event-free Survival
Description: Defined as time from randomization to the first documentation of event where events considered are 1) disease progression, per RECIST, prior to surgery, 2) surgery with R2 resection, 3) recurrent disease following surgery, or 4) death due to any cause. Will be estimated using the method of Kaplan-Meier in each arm and compared between treatment groups using the log-rank test. The correlation between pathologic complete response (pCR) status and event-free survival time will be assessed by Cox model with landmark approach.
Time Frame: 4 years and 7 months
Population: Excluded from analysis were 6 patients that withdrew or progressed prior to treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 (mFOLFIRINOX + Surgery + FOLFOX) | Arm 2 (mFOLFIRINOX + Radiation + Surgery + FOLFOXx)
Number analyzed (Participants) | 65 | 55
Months | 15.0 [11.2 to 21.9] | 10.2 [6.7 to 17.3]

4. Secondary Outcome: Pathologic Complete Rate (pCR) Rate
Description: Defined as the percentage of patients in whom a pCR was confirmed by histopathologic review of the surgical specimen. Chi-square test (or Fisher's exact test if the data in contingency table is sparse) will be used to compare pCR resection rate between two treatment arms. Sensitivity analysis will be conducted among patients in cohort 1) and cohort 2). The association between pCR rate and OS/progression free survival (PFS) will be assessed by log-rank test and Cox model.
Time Frame: 24 months
Population: Excluded from analysis were 6 patients that withdrew or progressed prior to treatment.
Measure: Number; unit: percentage of patients
Arm/Group | Arm 1 (mFOLFIRINOX + Surgery + FOLFOX) | Arm 2 (mFOLFIRINOX + Radiation + Surgery + FOLFOXx)
Number analyzed (Participants) | 65 | 55
percentage of patients | 0 | 11

5. Secondary Outcome: Incidence of Adverse Events Assessed Per Common Terminology Criteria for Adverse Events (CTCAE) Version 4 and the Patient-Reported Outcomes Version of the CTCAE
Description: Overall adverse event rates will be compared between treatment groups using Chi-square test (or Fisher's exact test if the data in contingency table is sparse).
Time Frame: 1 year
Population: All patients that were treated and assessed for adverse events
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (mFOLFIRINOX + Surgery + FOLFOX) | Arm 2 (mFOLFIRINOX + Radiation + Surgery + FOLFOXx)
Number analyzed (Participants) | 66 | 55
Participants | 66 | 55

ADVERSE EVENTS:
Time Frame: Adverse events and Serious Adverse events were collected for 2 years and all cause mortality was collected for 4 years and 7 months.
Arm/Group | Arm 1 (mFOLFIRINOX + Surgery + FOLFOX) | Arm 2 (mFOLFIRINOX + Radiation + Surgery + FOLFOXx)
All-Cause Mortality (participants affected / at risk) | 42/66 | 26/55
Serious Adverse Events (participants affected / at risk) | 33/66 | 28/55
Other Adverse Events (participants affected / at risk) | 64/66 | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (mFOLFIRINOX + Surgery + FOLFOX) (N=66) | Arm 2 (mFOLFIRINOX + Radiation + Surgery + FOLFOXx) (N=55)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (4)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 4 (6)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (8)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (4)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (6)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (3)
Chills (General disorders) | 1 (1) | 1 (1)
Death NOS (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (3)
Fever (General disorders) | 1 (1) | 3 (8)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 4 (4) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 3 (3) | 1 (2)
Infections and infestations - Oth spec (Infections and infestations) | 7 (7) | 3 (3)
Sepsis (Infections and infestations) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 6 (6) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
Weight loss (Investigations) | 0 (0) | 2 (2)
White blood cell decreased (Investigations) | 3 (3) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (3)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 3 (4) | 1 (2)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (mFOLFIRINOX + Surgery + FOLFOX) (N=66) | Arm 2 (mFOLFIRINOX + Radiation + Surgery + FOLFOXx) (N=55)
Anemia (Blood and lymphatic system disorders) | 35 (118) | 24 (112)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (8) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 2 (2)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 3 (5) | 2 (16)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Scleral disorder (Eye disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 18 (37) | 18 (36)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 5 (15) | 5 (26)
Constipation (Gastrointestinal disorders) | 16 (40) | 9 (10)
Diarrhea (Gastrointestinal disorders) | 56 (272) | 47 (191)
Dry mouth (Gastrointestinal disorders) | 9 (36) | 7 (27)
Dyspepsia (Gastrointestinal disorders) | 5 (10) | 5 (14)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 5 (10) | 6 (23)
Gastritis (Gastrointestinal disorders) | 1 (3) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 (16) | 5 (10)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 2 (3) | 3 (6)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (3)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 9 (16) | 12 (23)
Nausea (Gastrointestinal disorders) | 57 (279) | 46 (222)
Oral dysesthesia (Gastrointestinal disorders) | 3 (4) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 3 (4)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 18 (25) | 15 (35)
Chills (General disorders) | 2 (2) | 2 (3)
Edema limbs (General disorders) | 6 (11) | 6 (11)
Fatigue (General disorders) | 61 (395) | 52 (307)
Fever (General disorders) | 5 (6) | 3 (3)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Gen disord and admin site conds-Oth spec (General disorders) | 5 (29) | 1 (9)
Localized edema (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 2 (5) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (2)
Pain (General disorders) | 4 (9) | 8 (15)
Bile duct stenosis (Hepatobiliary disorders) | 5 (15) | 9 (40)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 (2) | 1 (3)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatic infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 2 (2) | 1 (1)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 3 (5) | 0 (0)
Skin infection (Infections and infestations) | 2 (3) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 4 (4) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (6) | 3 (3)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 26 (77) | 16 (51)
Alkaline phosphatase increased (Investigations) | 23 (78) | 19 (83)
Aspartate aminotransferase increased (Investigations) | 22 (53) | 14 (40)
Blood bilirubin increased (Investigations) | 15 (24) | 11 (13)
Creatinine increased (Investigations) | 3 (5) | 0 (0)
Investigations - Other, specify (Investigations) | 2 (2) | 1 (2)
Lymphocyte count decreased (Investigations) | 7 (10) | 7 (29)
Neutrophil count decreased (Investigations) | 16 (20) | 15 (20)
Platelet count decreased (Investigations) | 20 (54) | 20 (55)
Weight loss (Investigations) | 42 (162) | 33 (142)
White blood cell decreased (Investigations) | 12 (18) | 10 (16)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 23 (97) | 21 (86)
Dehydration (Metabolism and nutrition disorders) | 7 (11) | 8 (18)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 15 (40) | 9 (28)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 42 (157) | 34 (124)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (18) | 9 (21)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 21 (56) | 21 (43)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (29) | 7 (13)
Hyponatremia (Metabolism and nutrition disorders) | 10 (13) | 5 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (6) | 3 (3)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (14) | 5 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 6 (17) | 5 (15)
Dysarthria (Nervous system disorders) | 2 (5) | 3 (3)
Dysesthesia (Nervous system disorders) | 3 (18) | 2 (3)
Dysgeusia (Nervous system disorders) | 14 (40) | 14 (58)
Headache (Nervous system disorders) | 3 (10) | 5 (8)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (2)
Nervous system disorders - Oth spec (Nervous system disorders) | 2 (9) | 2 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (2)
Paresthesia (Nervous system disorders) | 6 (11) | 7 (26)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 49 (269) | 39 (215)
Somnolence (Nervous system disorders) | 0 (0) | 2 (3)
Anxiety (Psychiatric disorders) | 3 (9) | 4 (11)
Confusion (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 3 (9) | 2 (5)
Insomnia (Psychiatric disorders) | 3 (8) | 5 (8)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 2 (3)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (2)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 1 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 1 (4)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (2)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (20) | 6 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (8) | 1 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (46) | 7 (30)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (11) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (13) | 0 (0)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (6) | 3 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (17) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 2 (2)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 2 (4)
Hypertension (Vascular disorders) | 7 (28) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 4 (5)
Thromboembolic event (Vascular disorders) | 2 (3) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT02839343/Prot_SAP_000.pdf